CLINICAL TRIAL: NCT04011176
Title: Microcurrent Treatment for Chronic Debilitating Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Crawford (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Paul Crawford, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20190097h
Record Dates: First submitted 2019-07-02; First posted 2019-07-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain; Opioid Use
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard treatment + placebo (Placebo Comparator): Placing the microcurrent pads on the patient but not turning on the microcurrent box for 30 minutes once a week for 6 weeks
  Interventions: Procedure: Standard treatment + placebo
- Standard treatment + Microcurrent Therapy (Experimental): 100-300µA microcurrent delivered for 20-300 minutes, once a week for 6 weeks
  Interventions: Procedure: Standard treatment + Microcurrent Therapy

INTERVENTIONS:
Procedure: Standard treatment + placebo — Placebo microcurrent
  Arms: Standard treatment + placebo
Procedure: Standard treatment + Microcurrent Therapy — Actual microcurrent
  Arms: Standard treatment + Microcurrent Therapy

SUMMARY:
To compare the efficacy of standard pain treatment and placebo (a microcurrent faux treatment) as opposed to standard pain treatment and microcurrent therapy in any primary care patients over a three month period.

DETAILED DESCRIPTION:
This study is not intended to be definitive and should be considered an exploratory randomized trial to determine conditions for which microcurrent is more effective. Thus, extensive subgroup analyses will be performed so that definitive trials can be developed. This is a single-blind study where subjects will not know if they are receiving microcurrent treatment.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male and female Active Duty members and DoD beneficiaries
* Age 18 years or older
* Chronic debilitating pain
* PROMIS-57 T score is 60 or above

Exclusion Criteria:

* Pregnant
* Implanted pacemaker
* Spinal cord stimulator
* Illicit drug use including marijuana use
* Epilepsy or a history of seizures
* Other implanted device (e.g., insulin pump, opioid pump, or defibrillator)
* Chronic debilitating pain referred or recruited as measured by PROMIS-57 T score is below 60

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | PRE-TREATMENT: time 0 (week 0)
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). In most cases 50 equals the mean in the U.S. general population.
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | PRE-TREATMENT: time 1 (week 1)
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). In most cases 50 equals the mean in the U.S. general population.
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | PRE-TREATMENT: time 2 (week 2)
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). In most cases 50 equals the mean in the U.S. general population.
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | PRE-TREATMENT: time 3 (week 3)
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). In most cases 50 equals the mean in the U.S. general population.
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | PRE-TREATMENT: time 4 (week 4)
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). In most cases 50 equals the mean in the U.S. general population.
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | PRE-TREATMENT: time 5 (week 5)
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). In most cases 50 equals the mean in the U.S. general population.
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | PRE-TREATMENT: time 6 (week 12)
  PROMIS measures provide a common metric: the T-score (mean = 50, standard deviation = 10). In most cases 50 equals the mean in the U.S. general population.
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | POST-TREATMENT: time 0 (week 0)
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | POST-TREATMENT: time 1 (week 1)
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | POST-TREATMENT: time 2 (week 2)
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | POST-TREATMENT: time 3 (week 3)
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | POST-TREATMENT: time 4 (week 4)
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | POST-TREATMENT: time 5 (week 5)
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | POST-TREATMENT: time 6 (week 12)
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Patient-Reported Outcomes Information System (PROMIS) -57 Profile standardized T-Scores | SCREENING
  PROMIS-57 is a collection of 8-item short forms assessing anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities as well as a single pain intensity item.
Measure Yourself Medical Outcome Profile (MYMOP) | PRE-TREATMENT: time 0 (week 0)
  MYMOP measures the outcomes that the patient considers the most important.The patient chooses one or two symptoms that they are seeking help with, and that they consider to be the most important. They also choose an activity of daily living that is limited or prevented by this problem. These choices are written down in the patient's own words and the patient scores them for severity over the past week on a seven-point scale. Lastly wellbeing is scored on a similar scale.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | PRE-TREATMENT: time 1 (week 1)
  MYMOP measures the outcomes that the patient considers the most important.The patient chooses one or two symptoms that they are seeking help with, and that they consider to be the most important. They also choose an activity of daily living that is limited or prevented by this problem. These choices are written down in the patient's own words and the patient scores them for severity over the past week on a seven-point scale. Lastly wellbeing is scored on a similar scale.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | PRE-TREATMENT: time 2 (week 2)
  MYMOP measures the outcomes that the patient considers the most important.The patient chooses one or two symptoms that they are seeking help with, and that they consider to be the most important. They also choose an activity of daily living that is limited or prevented by this problem. These choices are written down in the patient's own words and the patient scores them for severity over the past week on a seven-point scale. Lastly wellbeing is scored on a similar scale.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | PRE-TREATMENT: time 3 (week 3)
  MYMOP measures the outcomes that the patient considers the most important.The patient chooses one or two symptoms that they are seeking help with, and that they consider to be the most important. They also choose an activity of daily living that is limited or prevented by this problem. These choices are written down in the patient's own words and the patient scores them for severity over the past week on a seven-point scale. Lastly wellbeing is scored on a similar scale.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | PRE-TREATMENT: time 4 (week 4)
  MYMOP measures the outcomes that the patient considers the most important.The patient chooses one or two symptoms that they are seeking help with, and that they consider to be the most important. They also choose an activity of daily living that is limited or prevented by this problem. These choices are written down in the patient's own words and the patient scores them for severity over the past week on a seven-point scale. Lastly wellbeing is scored on a similar scale.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | PRE-TREATMENT: time 5 (week 5)
  MYMOP measures the outcomes that the patient considers the most important.The patient chooses one or two symptoms that they are seeking help with, and that they consider to be the most important. They also choose an activity of daily living that is limited or prevented by this problem. These choices are written down in the patient's own words and the patient scores them for severity over the past week on a seven-point scale. Lastly wellbeing is scored on a similar scale.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | PRE-TREATMENT: time 6 (week 12)
  MYMOP measures the outcomes that the patient considers the most important.The patient chooses one or two symptoms that they are seeking help with, and that they consider to be the most important. They also choose an activity of daily living that is limited or prevented by this problem. These choices are written down in the patient's own words and the patient scores them for severity over the past week on a seven-point scale. Lastly wellbeing is scored on a similar scale.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | POST-TREATMENT: time 0 (week 0)
  MYMOP measures the outcomes that the patient considers the most important.On follow-up questionnaires the wording of the previously chosen items is unchanged.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | POST-TREATMENT: time 1 (week 1)
  MYMOP measures the outcomes that the patient considers the most important.On follow-up questionnaires the wording of the previously chosen items is unchanged.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | POST-TREATMENT: time 2 (week 2)
  MYMOP measures the outcomes that the patient considers the most important.On follow-up questionnaires the wording of the previously chosen items is unchanged.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | POST-TREATMENT: time 3 (week 3)
  MYMOP measures the outcomes that the patient considers the most important.On follow-up questionnaires the wording of the previously chosen items is unchanged.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | POST-TREATMENT: time 4 (week 4)
  MYMOP measures the outcomes that the patient considers the most important.On follow-up questionnaires the wording of the previously chosen items is unchanged.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | POST-TREATMENT: time 5 (week 5)
  MYMOP measures the outcomes that the patient considers the most important.On follow-up questionnaires the wording of the previously chosen items is unchanged.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Measure Yourself Medical Outcome Profile (MYMOP) | POST-TREATMENT: time 6 (week 12)
  MYMOP measures the outcomes that the patient considers the most important.On follow-up questionnaires the wording of the previously chosen items is unchanged.
  Produces a 7-point scale (0=as good as it could be, 6=as bad as it could be) for individual items of Symptoms, Activity, and Wellbeing as well as the MYMOP profile score
Defense and Veterans Pain Rating Scale (DVPRS) | PRE-TREATMENT: time 0 (week 0)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | PRE-TREATMENT: time 1 (week 1)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | PRE-TREATMENT: time 2 (week 2)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | PRE-TREATMENT: time 3 (week 3)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | PRE-TREATMENT: time 4 (week 4)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | PRE-TREATMENT: time 5 (week 5)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | PRE-TREATMENT: time 6 (week 6)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | POST-TREATMENT: time 0 (week 0)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | POST-TREATMENT: time 1 (week 1)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | POST-TREATMENT: time 2 (week 2)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | POST-TREATMENT: time 3 (week 3)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | POST-TREATMENT: time 4 (week 4)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | POST-TREATMENT: time 5 (week 5)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.
Defense and Veterans Pain Rating Scale (DVPRS) | POST-TREATMENT: time 6 (week 6)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VHA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used.

SECONDARY OUTCOMES:
Opioids taken | screening, time 0 (week 0), time 1 (week 1), time 2 (week 2), time 3 (week 3), time 4 (week 4), time 5 (week 5), time 6 (week 12)
  Opioids taken measured in morphine equivalent units (MEU; milligrams)

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

REFERENCES:
- [Background] Varney SM, Bebarta VS, Mannina LM, Ramos RG, Ganem VJ, Carey KR. Emergency medicine providers' opioid prescribing practices stratified by gender, age, and years in practice. World J Emerg Med. 2016;7(2):106-10. doi: 10.5847/wjem.j.1920-8642.2016.02.004. PMID 27313804
- [Background] Jeffery DD, Babeu LA, Nelson LE, Kloc M, Klette K. Prescription drug misuse among U.S. active duty military personnel: a secondary analysis of the 2008 DoD survey of health related behaviors. Mil Med. 2013 Feb;178(2):180-95. doi: 10.7205/milmed-d-12-00192. PMID 23495464
- [Background] Jeffery DD, May L, Luckey B, Balison BM, Klette KL. Use and abuse of prescribed opioids, central nervous system depressants, and stimulants among U.S. active duty military personnel in FY 2010. Mil Med. 2014 Oct;179(10):1141-8. doi: 10.7205/MILMED-D-14-00002. PMID 25269133
- [Background] Chen JH, Humphreys K, Shah NH, Lembke A. Distribution of Opioids by Different Types of Medicare Prescribers. JAMA Intern Med. 2016 Feb;176(2):259-61. doi: 10.1001/jamainternmed.2015.6662. No abstract available. PMID 26658497
- [Background] Levy B, Paulozzi L, Mack KA, Jones CM. Trends in Opioid Analgesic-Prescribing Rates by Specialty, U.S., 2007-2012. Am J Prev Med. 2015 Sep;49(3):409-13. doi: 10.1016/j.amepre.2015.02.020. Epub 2015 Apr 18. PMID 25896191
- [Background] Gabriel A, Sobota R, Gialich S, Maxwell GP. The use of Targeted MicroCurrent Therapy in postoperative pain management. Plast Surg Nurs. 2013 Jan-Mar;33(1):6-8; quiz 9-10. doi: 10.1097/PSN.0b013e3182844219. PMID 23446501
- [Background] Pilla A, Fitzsimmons R, Muehsam D, Wu J, Rohde C, Casper D. Electromagnetic fields as first messenger in biological signaling: Application to calmodulin-dependent signaling in tissue repair. Biochim Biophys Acta. 2011 Dec;1810(12):1236-45. doi: 10.1016/j.bbagen.2011.10.001. Epub 2011 Oct 8. PMID 22005645
- [Background] Rohde C, Chiang A, Adipoju O, Casper D, Pilla AA. Effects of pulsed electromagnetic fields on interleukin-1 beta and postoperative pain: a double-blind, placebo-controlled, pilot study in breast reduction patients. Plast Reconstr Surg. 2010 Jun;125(6):1620-1629. doi: 10.1097/PRS.0b013e3181c9f6d3. PMID 20527063
- [Background] Strauch B, Herman C, Dabb R, Ignarro LJ, Pilla AA. Evidence-based use of pulsed electromagnetic field therapy in clinical plastic surgery. Aesthet Surg J. 2009 Mar-Apr;29(2):135-43. doi: 10.1016/j.asj.2009.02.001. PMID 19371845
- [Background] Iodice P, Lessiani G, Franzone G, Pezzulo G. Efficacy of pulsed low-intensity electric neuromuscular stimulation in reducing pain and disability in patients with myofascial syndrome. J Biol Regul Homeost Agents. 2016 Apr-Jun;30(2):615-20. PMID 27358158
- [Background] Taylor AG, Anderson JG, Riedel SL, Lewis JE, Kinser PA, Bourguignon C. Cranial electrical stimulation improves symptoms and functional status in individuals with fibromyalgia. Pain Manag Nurs. 2013 Dec;14(4):327-335. doi: 10.1016/j.pmn.2011.07.002. Epub 2011 Oct 6. PMID 24315255
- [Background] Rajpurohit B, Khatri SM, Metgud D, Bagewadi A. Effectiveness of transcutaneous electrical nerve stimulation and microcurrent electrical nerve stimulation in bruxism associated with masticatory muscle pain--a comparative study. Indian J Dent Res. 2010 Jan-Mar;21(1):104-6. doi: 10.4103/0970-9290.62816. PMID 20427917
- [Background] Koopman JS, Vrinten DH, van Wijck AJ. Efficacy of microcurrent therapy in the treatment of chronic nonspecific back pain: a pilot study. Clin J Pain. 2009 Jul-Aug;25(6):495-9. doi: 10.1097/AJP.0b013e31819a6f3e. PMID 19542797